CLINICAL TRIAL: NCT05244395
Title: Development of a New Instrument to Evaluate Gait Characteristics of Individuals With Duchenne Muscular Dystrophy: Gait Assessment Scale for Duchenne Muscular Dystrophy, and Its Validity and Reliability
Brief Title: Development of a New Instrument to Evaluate Gait Characteristics of Individuals With Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güllü AYDIN YAĞCIOĞLU, Research Assistant, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GO 20/1058
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Duchenne Muscular Dystrophy; Gait Disorders in Children; Gait Disorders, Neurologic
Keywords: Duchenne Muscular Dystrophy; gait pattern; scale development; reliability and validity; gait analysis
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Duchenne Muscular Dystrophy Gait Assessment Scale (Experimental): The DMD-GAS was developed using the two-round Delphi method. After a detailed literature review, the items of scale were compiled. The DMD-GAS was designed to consist of 10 items and each item scored as 0,1,2. The DMD-GAS was presented to the expert group (10 physical therapists), who had experience in the management of patients with DMD. According to the scale items, it is classified as 2: no compensation, 1: minimal compensation, and 0: excessive compensation for the relevant body part.
  Interventions: Other: Duchenne Muscular Dystrophy Gait Assessment Scale

INTERVENTIONS:
Other: Duchenne Muscular Dystrophy Gait Assessment Scale — a special gait assessment scale for Duchenne Muscular Dystrophy patients

SUMMARY:
The aim of this study was to develop a gait assessment instrument for Duchenne Muscular Dystrophy patients (DMD-GAS), and investigate its validity and reliability.The scale was developed considering the expert opinions which included 10 physiotherapists who had experience in the management of patients with DMD over the 2-round Delphi method, and the Content Validity Index (CVI) was calculated. The final version of the DMD-GAS that was agreed upon the experts consisted of 10 items, and each item scored between 0 and 2. The intra-rater reliability was established by the video analysis of children with a 1-month interval and inter-rater reliability was determined by the scores of 3 physiotherapists. The criterion validity was determined by investigating the relationship between the total score of the DMD-GAS and Motor Function Measure (MFM), 6 Minute Walk Test (6MWT), and the data obtained from GAITRite system.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with DMD
2. Be between Levels I-V according to Brooke Lower Limb Extremity Functional Classification
3. Being between the ages of 5-18
4. Agreeing to participate in the research voluntarily

Exclusion Criteria:

1. Insufficient cooperation with the physiotherapist,
2. Have had any injury and/or surgery of the lower extremities in the last 6 months,
3. Having neurological problems in addition to DMD. -

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Duchenne Muscular Dystrophy Gait Assessment Scale (DMD-GAS) | 15-20 minutes
  The scale which developed specifically for DMD with this study. The DMD-GAS was designed to consist of 10 items and each item scored as 0 (excessive compensation in the relevant body part), 1 (minimal compensation) or 2 (no compensation). Low score indicate compensated gait.
Motor Function Measure (MFM) | 20-30 minutes
  MFM, which was valid and reliable in Neuromuscular Diseases, was used for gross motor function assessment. The items in MFM, which evaluate functions in 3 different sections (D1, standing position and transfers; D2, axial and proximal motor function; D3, distal motor function) in 32 items in total, are scored between 0-3. 0; cannot initiate any movement and maintain the starting position, 1; partially completes the exercise, 2; performs the exercise slowly and visibly clumsily, with compensations, 3; performs the exercise in the specified standard pattern. High scores indicate higher motor function and the result is expressed as a percentage of the maximum possible score to enable comparison with other scores

SECONDARY OUTCOMES:
6 meter walking test (6MWT) | 6 minutes
  6MWT is an assessment that was developed by Balke in the 1960s and has validity and reliability for DMD patients. The maximum distance that the patient can walk in 6 minutes is recorded as meters.

CONTACTS AND LOCATIONS:
Overall Officials: Güllü Aydın Yağcıoğlu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aydin Yagcioglu G, Alemdaroglu Gurbuz I, Topuz S, Yilmaz O. Development of a new instrument to evaluate gait characteristics of individuals with Duchenne Muscular Dystrophy: Gait Assessment Scale for Duchenne Muscular Dystrophy, and its validity and reliability. Early Hum Dev. 2023 Oct;185:105843. doi: 10.1016/j.earlhumdev.2023.105843. Epub 2023 Aug 23. PMID 37672897